CLINICAL TRIAL: NCT06280898
Title: Analysis of Perioperative Factors Affecting Early Postoperative Kidney Graft Function Recovery in Patients Undergoing Living Kidney Transplant Surgery
Brief Title: Perioperative Factors and Early Postoperative Kidney Graft Function Recovery
Status: Completed | Type: Observational
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Min Suk Chae, Professor, Seoul St. Mary's Hospital
Other Study IDs: KC22RISI0395
Record Dates: First submitted 2024-02-16; First posted 2024-02-28 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Heart Injuries; Kidney Transplant; Complications
MeSH Terms: conditions — Heart Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- nonischemic
- ischemic
  Interventions: Procedure: Remote ischemic conditioning

INTERVENTIONS:
Procedure: Remote ischemic conditioning — Remote ischemic condition
  Groups: ischemic

SUMMARY:
Divided into two groups based on acute kidney injury: non-acute kidney injury group vs. non-acute kidney injury group. Acute kidney injury group, Acute Kidney Injury Network (AKIN), Risk, Injury, Failure, Loss of kidney function, and End-stage kidney disease (RIFLE), or Kidney Disease: Improving Global Outcomes (KDIGO) I would like to divide it according to the definition. After testing the normal distribution of patients, donors, grafts, types of immunosuppressants, surgery/anesthesia factors, and blood test findings between the two groups through the Shapiro-Wilk test, continuous data was tested using the student t-test or Mann-Whitney U test. Sizes are compared using , and categorical data is compared with proportions using the χ2 test or Fisher's exact test. Analysis of factors related to acute kidney injury will be performed through univariate and multivariate logistic regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 19 years or older who underwent kidney transplant surgery in the operating room

Exclusion Criteria:

* Pediatric patients under 19 years of age
* Patients with multiple organ transplants, including kidney transplants
* Patients undergoing re-kidney transplant surgery
* Patient examination findings missing from electronic medical record

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 19 or older who underwent kidney transplant surgery in the operating room of Seoul St. Mary's Hospital from January 1, 2016 to March 28, 2022.
Sampling Method: Probability Sample
Enrollment: 539 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-03-14 (Actual)

PRIMARY OUTCOMES:
Troponin I | up to 24 hour postoperatively
  Troponin I difference in two groups

SECONDARY OUTCOMES:
Troponin T | up to 24 hour postoperatively
  Troponin T difference in two groups
QTc interval | up to 24 hour postoperatively
  OTc interval difference in two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul St. Mary's hospital, Seoul, South Korea